CLINICAL TRIAL: NCT04162665
Title: Pre-operative Adaptive Short Course Radiation Therapy in Gastric Cancer
Brief Title: Pre-operative Adaptive Short Court Radiation Therapy in Gastric Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual and funding sponsor declared bankruptcy.
Sponsor: Washington University School of Medicine (Other)
Collaborators: Viewray Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201911059
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Gastric Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Pre-operative adaptive short course radiation therapy (Experimental): Consenting and eligible patients will receive adaptive short course radiation therapy (SCRT) (25 Gy at in 5 fractions), followed by standard of care total neoadjuvant chemotherapy followed by standard of care gastrectomy or esophagogastrectomy. The recommended SOC chemotherapy options are CAPOX, FOLFOX, or FLOT, but any SOC total neoadjuvant chemotherapy may be given at the discretion of the treating medical oncologist after consultation with the study chair. Patients who are not able to complete their full total neoadjuvant therapy regimen prior to surgery may complete chemotherapy postoperatively at the discretion of the treating physician.
  Interventions: Radiation: Adaptive short course radiation therapy; Drug: Standard of care chemotherapy regimen

INTERVENTIONS:
Radiation: Adaptive short course radiation therapy — Radiation must be livered with adaptive planning and MR gating or CBCT breath hold treatment.
Drug: Standard of care chemotherapy regimen — The recommendations are CAPOX, FOLFOX, or FLT.

SUMMARY:
Gastric cancer is a global health issue as the world's fifth most common malignancy and third leading cause of cancer mortality, respectively. Preoperative radiation therapy may improve overall survival (OS) but is seldom used. There is precedent for preoperative chemoradiation, as it is the standard of care for esophageal and gastroesophageal junction tumors. However, reluctance of physicians to prescribe preoperative radiation therapy in gastric cancer may be due to the large treatment fields necessary to account for stomach motion. Adaptive radiation therapy may permit decreased field sizes and more accurate dose delivery. In traditional CT based radiation delivery the same radiation plan is delivered each day without assessment of inter-fraction or intra-fraction motion. Adaptive radiation therapy permits the physician to contour the unique anatomy daily to generate a new plan to account for day to day organ motion. Real-time MR imaging is also used during the treatment so that radiation is only delivered when the tumor is within the pre-specified target area. Thus, adaptive radiation therapy may overcome traditional barriers of radiation delivery in gastric cancer and improve oncologic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed histologically or cytologically gastric adenocarcinoma. (Siewert III acceptable: the bulk of tumor should be in stomach; gastric tumors with extension to the gastroesophageal junction are permitted.) Patients with T1-3N0-2 are eligible. Patients with N3, or T4 disease are not eligible.
* Known T-stage defined by EUS. Must have had CT of the chest/abdomen/pelvis with contrast.
* Medically eligible to receive standard of care chemotherapy.
* At least 19 years of age
* ECOG performance status ≤ 2

Normal bone marrow and organ function as defined below:

* Absolute neutrophil count ≥ 1,500 cells/mm3
* Platelets ≥ 100,000 cells/mm3
* Creatinine clearance > 50 mL/min

  * The effects of the various chemotherapy agents used in this study on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of the study, and one month after completion of the study
  * Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Prior surgery, radiation, or chemotherapy for gastric or esophageal cancer.
* Prior surgery to the esophagus or stomach that would alter the radiation treatment field or stomach motion.
* Siewert I-II GE junction tumor
* Any active malignancy within 2 years of enrollment that may alter the course of gastric cancer. (Apparently cured localized malignancy or advanced, but indolent malignancy with significantly more favorable prognosis are allowed).
* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to chemotherapeutic agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, diabetes, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia that are considered clinically significant as determined by the treating physician.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended. Recommend exclusion of specific ART agents based on predicted drug-drug interactions (i.e. for sensitive CYP3A4 substrates, concurrent strong CYP3A4 inhibitors (ritonavir and cobicistat) or inducers (efavirenz) should be contraindicated).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2024-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Kim, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the journal publication, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending ending 36 months following publication
Access Criteria: Investigators whose proposed use of the data has been approved by the Washington University School of Medicine IRB. The data will be available for individual participant data meta-analysis. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pre-operative Adaptive Short Course Radiation Therapy
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pre-operative Adaptive Short Course Radiation Therapy
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 73.5 [60 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Complete Pathologic Response (pCR - Primary and Nodal) Rate
Description: pCR: no pathological signs of cancer
Time Frame: At the time of surgery (approximately 4.5 months)
Population: 2 participants did not have surgery due to poor functional status and were not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-operative Adaptive Short Course Radiation Therapy
Number analyzed (Participants) | 2
Participants | 2

2. Secondary Outcome: Number of Participants With Local Control
Description: Local control calculated from start of radiation.
Time Frame: At 1 year post radiation
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-operative Adaptive Short Course Radiation Therapy
Number analyzed (Participants) | 4
Participants | 4

3. Secondary Outcome: Number of Grade 3 or Greater Toxicity as Defined by CTCAE Version 5.0
Time Frame: From baseline through 12 months after surgery/definitive end of treatment (estimated to be 16.5 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-operative Adaptive Short Course Radiation Therapy
Number analyzed (Participants) | 4
Participants
  Febrile neutropenia | 2
  Anemia | 2
  GI bleed | 1
  Gastric obstruction | 1
  Failure to thrive | 2
  Cholecystitis | 1
  Lung infection | 1
  Urinary tract infection | 1
  Blood bilirubin increased | 1
  Lymphocyte count decreased | 2
  Neutrophil count decreased | 1
  White blood cell decreased | 2
  Dehydration | 1
  Hypoalbuminemia | 2
  Syncope | 1
  Delirium | 1
  Pre-renal azotemia | 1
  Acute kidney injury | 1
  Percutaneous endoscopic gastromy tube clogging | 1

4. Secondary Outcome: Overall Survival
Description: -Overall survival from start of radiation.
Time Frame: At 1 year post radiation
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-operative Adaptive Short Course Radiation Therapy
Number analyzed (Participants) | 4
Participants | 4

5. Secondary Outcome: Number of Participants With Disease-free Survival
Description: -Disease free means no locoregional and distant recurrence
Time Frame: At 1 year post radiation
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-operative Adaptive Short Course Radiation Therapy
Number analyzed (Participants) | 4
Participants | 4

6. Secondary Outcome: Number of Patients Able to Complete a Full Course of Total Neoadjuvant Chemotherapy
Time Frame: Through completion of neoadjuvant chemotherapy (estimated to be 4.5 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-operative Adaptive Short Course Radiation Therapy
Number analyzed (Participants) | 4
Participants | 3

7. Other Pre Specified Outcome: Average Percentage Difference in Dose to Nearby Organs at Risk (OARs) Due to Variation in OAR Position
Time Frame: Completion of radiation therapy (up to 2 weeks)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Average Percent Difference in Coverage of Planning Target Volume (PTV) by 95% Isodose Line
Time Frame: Completion of radiation therapy (up to 2 weeks)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events and all-cause mortality was to be collected from baseline up to 12 months after surgery (or, for patients who do not undergo surgery, up to 12 months after definitive end of treatment).
Arm/Group | Pre-operative Adaptive Short Course Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-operative Adaptive Short Course Radiation Therapy (N=4)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
GI bleed (Gastrointestinal disorders) | 1
Gastric obstruction (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Pre-renal azotemia (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-operative Adaptive Short Course Radiation Therapy (N=4)
Anemia (Blood and lymphatic system disorders) | 2
Cytopenia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 3
Mouth sores (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Cold sensitivity (General disorders) | 1
Decreased appetite (General disorders) | 1
Edema limbs (General disorders) | 1
Failure to thrive (General disorders) | 1
Fatigue (General disorders) | 4
Bile duct stenosis (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
COVID-19 infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 2
Pancytopenia (Investigations) | 1
Platelet count decreased (Investigations) | 3
Vitamin D deficiency (Investigations) | 1
White blood cell decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 1
Electrolyte abnormality (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypovolemic hyponatremia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 3
Encephalopathy (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Altered mental status (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Percutaneous endoscopic gastromy tube clogging (Surgical and medical procedures) | 1
Hypotension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Due to the limited number of participants treated, the statistical analyses as stated in the protocol could not be performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/65/NCT04162665/Prot_SAP_000.pdf